CLINICAL TRIAL: NCT00685997
Title: Whole-body MR Imaging for Staging Malignant Lymphomas
Brief Title: Whole-body Magnetic Resonance Imaging (MRI) for Staging Malignant Lymphomas
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, R.A.J. Nievelstein, M.D., Ph.D., UMC Utrecht
Other Study IDs: 80-82310-98-08012
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Malignant Lymphoma; Hodgkin's Disease; Non-Hodgkin's Lymphoma
Keywords: Malignant lymphoma; Hodgkin's disease; Non-Hodgkin's lymphoma; Imaging; Whole-Body MRI; CT; Radiation
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Background:

The malignant lymphomas, Hodgkin´s disease (HD) and non-Hodgkin´s lymphoma (NHL), comprise approximately 5-6% of all malignancies in adults and account for 10% of childhood cancers. Once the diagnosis has been established histologically, extent of disease (staging) and response to therapy will be assessed by means of a computed tomography (CT) scan of the body. The staging at presentation is important for determining prognosis and choice of treatment. Unfortunately, CT is accompanied by a significant amount of radiation exposure which may induce second cancers. This is especially important in childhood, because rapidly dividing cells are more sensitive to radiation induced effects and children will have more years ahead in which cancerous changes might occur. New magnetic resonance imaging (MRI) techniques offer an alternative way for staging and follow-up of cancers, including the malignant lymphomas. Whole-body MRI (WB-MRI) is a radiation-free method which allows imaging of the body with excellent soft tissue contrast in a single examination.

Purpose:

The aim of this study is to examine if WB-MRI can replace CT in staging of patients with a malignant lymphoma.

Design:

This will be a multicenter, prospective, diagnostic cohort study (timeschedule: 36 months). 135 eligible patients will undergo WB-MRI on top of the protocolar imaging routinely done.

Study population:

Patients aged 8 years and older with a histological diagnosis of HD or NHL.

Statistical analysis:

The challenge of this study will be to show non-inferiority of WB-MRI compared to CT in staging malignant lymphoma. Testing of this hypothesis will be one-sided and performed using recently proposed techniques by Lui et al.

Radiation-related risk assessment:

A risk model will be used, based on the BEIR VII report, for modelling the late-term mortality from radiation induced tumors after exposure to ionizing radiation.

Economic evaluation:

Actual costs (from a societal perspective) will be determined for the two diagnostic tests. In case of clinical equivalence and similar costs or cost savings associated with MRI the latter can be considered dominant, obviating further economic evaluation. Otherwise, through modelling of expected long term health impact and associated outcomes such as quality of life and costs the incremental cost effectiveness will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients
* age: 8 years and older
* histologically proven Hodgkin's disease or non-Hodgkin's lymphoma
* patients scheduled for a CT of the body for initial staging
* participant's parents (participant < 18 years) or the participant (participant >18 years) must willingly give written informed consent prior to the start of the study
* whole-body MRI has to be performed within 10 days before or after CT, and before therapy has been started.

Exclusion Criteria:

* patients with a general contraindication for MRI (including cardiovascular pacemakers, claustrophobia)
* patients who have had a previous malignancy
* patients who are pregnant or nursing
* patients in whom therapy has already started after CT and before MRI could be performed

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients, aged 8 years and older, with newly diagnosed Hodgkin's disease or non-Hodgkin's lymphoma, who will undergo computed tomography (CT) for staging
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2008-06; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the clinical stage according to WB-MRI findings and according to CT-findings. This clinical stage will be determined according to the Ann Arbor classification system. | December 2010

SECONDARY OUTCOMES:
The secondary outcome will be a (subjective) assessment of image quality and presence of artefacts, for both T1-weighted and T2-weighted MR images as well as CT. | December 2010

CONTACTS AND LOCATIONS:
Overall Officials: Rutger A. J. Nievelstein, MD PhD, Principal Investigator — UMC Utrecht
Locations (3):
- Netherlands (3):
  - Academic Medical Center Amsterdam, Amsterdam, North Holland
  - Meander Medical Center Amersfoort, Amersfoort, Utrecht
  - University Medical Center Utrecht, Utrecht, Utrecht

REFERENCES:
- [Background] Brennan DD, Gleeson T, Coate LE, Cronin C, Carney D, Eustace SJ. A comparison of whole-body MRI and CT for the staging of lymphoma. AJR Am J Roentgenol. 2005 Sep;185(3):711-6. doi: 10.2214/ajr.185.3.01850711. PMID 16120924
- [Background] Kellenberger CJ, Epelman M, Miller SF, Babyn PS. Fast STIR whole-body MR imaging in children. Radiographics. 2004 Sep-Oct;24(5):1317-30. doi: 10.1148/rg.245045048. PMID 15371611
- [Background] Lauenstein TC, Goehde SC, Herborn CU, Goyen M, Oberhoff C, Debatin JF, Ruehm SG, Barkhausen J. Whole-body MR imaging: evaluation of patients for metastases. Radiology. 2004 Oct;233(1):139-48. doi: 10.1148/radiol.2331030777. Epub 2004 Aug 18. PMID 15317952
- [Background] Antoch G, Vogt FM, Freudenberg LS, Nazaradeh F, Goehde SC, Barkhausen J, Dahmen G, Bockisch A, Debatin JF, Ruehm SG. Whole-body dual-modality PET/CT and whole-body MRI for tumor staging in oncology. JAMA. 2003 Dec 24;290(24):3199-206. doi: 10.1001/jama.290.24.3199. PMID 14693872
- [Background] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031